CLINICAL TRIAL: NCT02900872
Title: Systematic Chart Review of Carotidynia Patients
Acronym: TIPIC
Status: Completed | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: NI_ALR_2015_3
Record Dates: First submitted 2016-09-06; First posted 2016-09-14 (Estimated); Last update posted 2016-09-14 (Estimated); Status verified 2016-09

CONDITIONS: Carotidynia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective

SUMMARY:
Systematic retrospective study of medical charts and medical imaging files, of patients consulting for acute neck pain and presenting unclassified abnormalities on dedicated vessel imaging.

ELIGIBILITY:
Inclusion Criteria:

* acute cervical tenderness or neck pain fulfilling the characteristics of an idiopathic neck pain syndrome as defined by the International Headache Society in 1988
* the performing of a diagnostic imaging like MRI, CT or US of the cervical area with a dedicated vessel analysis
* unilateral or bilateral abnormalities of common carotid, carotid bifurcation or internal carotid arteries on dedicated vessel imaging.

Exclusion Criteria:

* patients without imaging, or without dedicated vessel analysis
* patients presenting with pain caused by a clearly identified vascular disease on dedicated vessel analysis imaging such as carotid occlusion, carotid dissection, vasculitis like giant cell arteritis.
* patients with no abnormality on cervical or vessel imaging

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult patients suffering from acute cervical pain or tenderness, fulfilling the characteristics of an idiopathic neck pain syndrome, and presenting with abnormalities of carotid arteries on dedicated vessel imaging
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2009-01; Primary Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Presence or absence of perivascular carotid artery enlargement on dedicated vessel imaging | Within 1 week following admission